CLINICAL TRIAL: NCT00477997
Title: The Effect of a Physiological Bolus of Growth Hormone (GH) on Insulin Signaling Pathways in Muscle Tissue From Healthy Adults
Brief Title: Effect of Growth Hormone on Insulin Signaling in Muscle Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Jens Otto Lunde Jørgensen, Aarhus University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: MM-GH-20070052
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Insulin Resistance
Keywords: Growth Hormone; Insulin Signaling; GH signaling
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Saline bolus + OGTT
  Interventions: Device: Physiological Bolus of Growth Hormone
- 2 (Other): GH-bolus and OGTT
  Interventions: Device: Physiological Bolus of Growth Hormone
- 3 (Other): GH-bolus
  Interventions: Device: Physiological Bolus of Growth Hormone

INTERVENTIONS:
Device: Physiological Bolus of Growth Hormone — 0,5 mg Norditropin

SUMMARY:
The purpose of this study is to examine the effects of a physiological bolus of growth hormone on insulin signaling pathways in muscle tissue in healthy lean men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Age between 18 and 30 years
* BMI ≤ 26

Exclusion Criteria:

* Known present disease including diabetes mellitus
* BMI > 26
* Uses any medication
* Consumes > 21 units of alcohol per week

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PI3-kinase activity i muscle tissue | 2 hours

SECONDARY OUTCOMES:
Growth Hormone Signaling Proteins in Muscle Tissue and other Insulin Signaling Proteins in Muscle Tissue | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, MD, DMSc, Principal Investigator — Department M (endocrinology and diabetes), Aarhus University Hospital, Norrebrogade 44, 8000 Aarhus C, Denmark
Locations (1):
- Department M (endocrinology and diabetes), Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Krusenstjerna-Hafstrom T, Madsen M, Vendelbo MH, Pedersen SB, Christiansen JS, Moller N, Jessen N, Jorgensen JO. Insulin and GH signaling in human skeletal muscle in vivo following exogenous GH exposure: impact of an oral glucose load. PLoS One. 2011 May 3;6(5):e19392. doi: 10.1371/journal.pone.0019392. PMID 21559284